CLINICAL TRIAL: NCT06545591
Title: Soluble Soluble Triggering Receptors Expressed on Myeloid Cells (sTREM) Predict Outcomes in Stroke Patients Receiving Endovascular Thrombectomy
Brief Title: Predictive Role of sTREM in Endovascular Thrombectomy Outcomes
Status: Recruiting | Type: Observational
Sponsor: The Affiliated Hospital of Xuzhou Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: XYFY2024-KL335-01
Record Dates: First submitted 2024-08-04; First posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Acute Ischemic Stroke
Keywords: Thrombectomy; soluble TREM-1; soluble TREM-2
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- EVT-stroke group: Patients with ischemic stroke who received endovascular thrombectomy (EVT) treatment
- non--EVT stroke group: The non--EVT stroke group was composed of patients with ischemic stroke without endovascular thrombectomy (EVT) treatment during the same period
- non--stroke control group: The non--stroke control group was composed of randomly selected stroke--free, age--matched and sex--matched individuals recruited from the health examination center.

SUMMARY:
Soluble triggering receptor expressed on myeloid cells (sTREM), which reflects microglia activation, has been reported closely associated with neuronal injury and neuroinflammation. This study is to investigatethe prognostic roles of sTREM (sTREM1 and sTREM2) in patients with ischemic stroke who underwent endovascular thrombectomy (EVT).

DETAILED DESCRIPTION:
For acute ischemic stroke, the current treatment strategy involves timely recanalization by intravenous thrombolysis and endovascular thrombectomy (EVT). Patients receiving EVT are more likely to achieve successful revascularization and long--term functional independence compared with those receiving standard medical treatment.1 In patients receiving EVT, significant predictors of a favorable functional outcome include minor initial stroke severity, successful recanalization, and shorter onset--to--treatment time. However, unfavorable outcomes can occur even after early successful recanalization in some cases.Triggering receptors expressed on myeloid cells (TREM-1 and TREM-2) are a familyof receptors involved in the immune system expressed on a variety of innate cells of the myeloid lineage, including microglia. sTREM, which reflects microglia activation, has been reported closely associated with neuronal injury and neuroinflammation. We enrolled adult patients with stroke who received EVT, with blood sampling immediately before (T1) and after EVT (T2), and at 24 hours after EVT (T3). Non--stroke controls and patients with non--EVT stroke were also enrolled. The plasma concentration of sTREM1 and sTREM2 were analyzed by ELISA. The medical information, image findings and levels of plasma sTREM1 and sTREM2 were analyzed to clarify the association with poor functional outcome (modified Rankin Scale 4-6) at 3 months after stroke.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 18 years old.
* Patients with acute large vessel occlusion within 24 hours of onset who will receive endovascular treatment.

Exclusion Criteria:

* Impossibility of getting a blood sample.
* Impossibility of performing the test (Invalid results).
* Refusal to provide the informed consent by the patient/relative.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: There will be 200 patients with stroke who underwent EVT (Endovascular Therapy), 50 patients with non--EVT stroke and 50 non--stroke controls.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Dynamic changes in plasma levels of sTREM-1 and sTREM-2 following Endovascular Therapy | From baseline to immediately, 24 hours, 3 days, and 7 days after Endovascular Therapy
  Plasma levels of sTREM-1 and sTREM-2 will be quantified using the ELISA method.

SECONDARY OUTCOMES:
favourable functional outcome, defined as modified Rankin Scale (mRS) 0-2 | 90 days
  mRS ranges from 0-6, high score means poor outcome
excellent functional outcome, defined as modified Rankin Scale (mRS) 0-1 | 30 days
  mRS ranges from 0-6, high score means poor outcome
early neurological improvement, defined as 4 or more decrease in National Institute of Health stroke scale (NIHSS) | 24 hours
  NIHSS ranges from 0-22, with high score meaning severe neurological deficit.
Hemorrhagic transformation | 72 hours
  Hemorrhagic transformation was diagnosed by Computed tomographic scans usually performed 24 to 72 hours after the procedure.Symptomatic intracranial hemorrhage was defined as neurologic deterioration (an increase of 4 or more points in the score on the NIHSS) and evidence of intracranial hemorrhage on imaging studies.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Neurology, Xuzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No